CLINICAL TRIAL: NCT04557111
Title: Quality and Satisfaction in CIED Remote Monitoring
Brief Title: Remote Care for CIED Patients in Korea
Status: Completed | Type: Observational
Sponsor: Saint Vincent's Hospital, Korea (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Principal Investigator, You Mi Hwang, Assistant Professor in Internal Medicine, Cardiology, Cardiac Electrophysiologist, Saint Vincent's Hospital, Korea
Other Study IDs: Remote Care Study
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Arrhythmias, Cardiac
Keywords: pacemaker; Implantable Cardioverter Defbrillator; Cardiac resynchronization therapy
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: remote monitoring — CIED monitoiring with remote monitoring device

SUMMARY:
This trial is for monitoring the quality and satisfaction of CIED patients who are naive with remote device monitoring.

DETAILED DESCRIPTION:
Patient satisfaction (using questionnaire) before and after wireless/wired monitoring and outpatient treatment time, variables in heart transplantation devices for wireless/wired monitoring, presence of heart failure, cardiovascular events such as arrhythmia, myocardial infarction or cerebral infarction, thromboembolism and admission related to cardiovascular cause. The questionnaire was adopted and modified from modified Korean version of HoMASQ (by YouMi Hwang,2021 from HoMASQ; Europace (2010))

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Biotronic CIED implanted in St. Vincent's Hospital, Catholic University of Korea, Republic of Korea
2. Patients who are literate and have perceptibility on questionnaire
3. Patients who followed up more than 6 months after CIED implantation
4. Patients with age of >20 years

Exclusion Criteria:

1. Patients with < 2 outpatient clinic visits during >6 months
2. Illiterate patients or inapprehensive of questionnaire
3. Patients with life expectancy of <1 year

Ages: 20 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes Biotronic CIED implanted patients in St. Vincent's Hospital, Catholic University of Korea, Republic of Korea. Study population are included if they are more than 20year old, followed up at outpatient clinic > 6 months after CIED implantation, and are literate and have perceptibility on questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction measurement before and after remote monitoring | 1 year
  Satisfaction measurement by questionnaire: Survey on telehealth patient experience(modified Korean version by YouMi Hwang,2020 from Bas-Villalobos, Form I) and Post remote monitoring satisfaction questionnaire, modified Korean version by YouMi Hwang,2020 from HoMASQ (Home Monitoring Acceptance and Satisfaction Questionnaire, Form II): Usually higher scores mean a worse outcome

SECONDARY OUTCOMES:
Any changes in prescription or patient visit schedule | 1 year
  Any changes in prescription or patient visit schedule based on remote monitoring
Out patient clinic time consumption per patient | 1 year
  Out patient clinic time consumption per patient
Changes in CIED parameters | 1 year
  Changes in CIED parameters during remote monitoring
Any cardiocerebrovascular events, deaths | 1 year
  Any cardiocerebrovascular events, deaths
Admission for heart failure or any cardiovascular intervention | 1 year
  Admission for heart failure or any cardiovascular intervention

CONTACTS AND LOCATIONS:
Overall Officials: YouMi Hwang, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- St. Vincent's Hospital, Suwon, Kyonggi Do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided